CLINICAL TRIAL: NCT05986747
Title: Feasibility and Acceptability Trial of a Video Based CBT Guided Self Help Intervention for People With no or Low Literacy: A Study From a Lower Middle-income Country.
Brief Title: Feasibility and Acceptability Trial of a Video Based CBT Guided Self Help Intervention for People With Low Literacy
Acronym: VCBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pakistan Association of Cognitive Therapists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PACTvCBT
Record Dates: First submitted 2023-06-23; First posted 2023-08-14 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Depression; Anxiety
Keywords: CBT; Self-help intervention; anxiety, depression; RCT
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants who met inclusion criteria will be randomly allocated to one of the groups, i.e. CBT video plus TAU (intervention group) or waitlist plus TAU (control group) in a 1:1 ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In the experimental group Video based CBT guided self help intervention will be provided
  Interventions: Behavioral: Video-based CBT guided self-help Interventions
- Control Group (No Intervention): In the control group, the patients screened for depression or anxiety received treatment as usual (TAU). TAU consisted of standard care under the responsible family physician. TAU in Pakistan largely consists of pharmacological treatment with anti-depressant medication and follow-up in an outpatient clinic.

INTERVENTIONS:
Behavioral: Video-based CBT guided self-help Interventions — Seven modules were developed from the corresponding modules of self help. Each video was of 3-5 minutes duration. Each week 2-3 videos will be sent to participants through secure WhatsApp connection. Participants received daily reminders in the form of short pre-recorded audio messages through whatsapp.
  Trained RAs will provide guidance as well as technical assistance during the intervention period. They will call participants once a week for 15 minutes. This call will include, feedback from previous session, explanation of current week and discussion on home work assignments.
  Arms: Experimental Group

SUMMARY:
This study aimed to assess the feasibility, acceptability, and preliminary efficacy of a video-based CBT guided self-help intervention 'Khushi or Khatoon' to treat anxiety and depression.

DETAILED DESCRIPTION:
Cognitive Behaviour Therapy (CBT) is now included in the National Treatment Guidelines in the UK. However, little progress has been made in its delivery in developing countries. Limited resources for the delivery of services and their concentration in big cities have implications for the choice of mode of delivery of treatment. A range of methods are needed to deliver treatment starting from self-help to more specialist interventions. Various CBT based self-help materials have been assessed and shown to be effective in the West . The effectiveness of a Culturally adapted CBT (CaCBT) based guided self-help has been reported, supervised by carers, against care as usual in patients with depression, who attend secondary care in Pakistan .

However, CBT requires a person to be literate, especially for guided self-help or self-help. Pakistan has a literacy rate (ability to read or write) of 58%. An estimated 67% of children study up to primary level (years 1-5) and an estimated 43% have achieved secondary education (up to year 12). These are mostly people from low socio-economic backgrounds who are less likely to suffer from mental health problems such as depression and anxiety. In order to overcome this barrier a video intervention based on self-help intervention is developed. This study aims at testing the feasibility, acceptability and preliminary effectiveness of this intervention.

This will be a rater-blind RCT to evaluate the feasibility and acceptability of video-based guided self-help in addition to treatment as usual (TAU) compared with the waitlist and TAU in Pakistan. This study will employ a pre-post measure and parallel design. It will be conducted from March 2023 to August 2023. Participants who met the inclusion criteria will be randomly allocated to one of the groups, i.e. CBT video plus TAU (intervention group) or waitlist plus TAU (control group) in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 to 65 years
2. without schooling
3. able to use a smartphone
4. Owning a smartphone or a personal computer with a reliable internet connection
5. Score of 8 or higher on Hospital Anxiety and Depression Scale-Depression or Anxiety Scales

Exclusion Criteria:

1. Substance use disorder according to DSM-5 criteria as determined by primary care clinician
2. Significant cognitive impairment (for example, profound learning disability or dementia) as determined by primary care clinician
3. Active psychosis as determined by their primary care clinician

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-11-28 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability trial of a video based CBT guided self-help intervention. | 12 weeks
  Feasibility and acceptability will be assessed through trial procedure, recruitment, retention and informal feedback from participants. Additionally clients satisfaction scale will be used to gather information on acceptability. At the end of the intervention, participants will be asked by RAs to describe their experience. They will be asked about to name the sessions that they found the most helpful or unhelpful, and to provide suggestions to improve the intervention. Those participants who completed less than five of seven modules will be considered drop-outs.

SECONDARY OUTCOMES:
Clinical Measures | 12 weeks
  The Hospital Anxiety and Depression Scale (HADS) will be used to measure Anxiety and Depression. The HADS is a rating scale consisting of 14 items, Each of the items is scored on a 4-point Likert scale from 0 (not present) to 3 (considerable). The sum of the individual items provides subscale scores on the HADS-D and the HADS-A, which may range between 0 and 21. A cut-off point of ≥8 for each of the constituent subscales is used to indicate probable caseness.
Functioning and Disability | 12 weeks
  The WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) will measure the functioning and disability. It covers 6 Domains of Functioning. the scores assigned to each of the items - "none" (0), "mild" (1) "moderate" (2), "severe" (3) and "extreme" (4) - are summed.

CONTACTS AND LOCATIONS:
Overall Officials: Farooq Naeem, Principal Investigator — PACT
Locations (1):
- Pakistan Association of Cognitive Therapists, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No